CLINICAL TRIAL: NCT05192785
Title: The Effects on Arterial Blood Gas, Venous Oxygen Saturation and Vital Findings of Incentive Spirometry Use With Inspiration and Expiration Techniques in Coronary Artery Bypass Surgery
Brief Title: The Effects Incentive Spirometry Use in Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Esma Gökçe, Principal Investigator (MSc), Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 50202081
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Incentive Spirometry; Oxygen Saturation
Keywords: Vital Signs; Coronary Heart Disease; Post-operative Care; Practice Nursing; Respiratory Nursing; Surgical Nursing
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group, patients who met the sampling criteria filled out the Consent and Information Forms with the researcher, and the breathing and coughing exercises, and early mobilization and pain control practices that were part of the routine clinical procedure were continued.
  Arterial and venous oxygen saturation values and vital signs were measured and recorded at the end of the first, second and third postoperative days on the Application Information form. The researchers and clinic nurses were responsible for the execution of applications and the follow-up and monitoring of the pulmonary rehabilitation care throughout the hospitalization of the patient.
- Incentive Spirometry Group (Experimental): The patients who met the sampling criteria were given consent and information forms in the preoperative period from their admission to the clinic by the researcher and the incentive spirometry (IS) application along with respiratory and cough exercises was explained, demonstrated and performed.
  In addition, all postoperative patients underwent a pain assessment using the visual analogue scale (VAS) pain scale every 4-6 hours every day prior to incentive spirometry implementation, and pain control was provided based on the results (with paracetamol and opioids in the clinical routine). The patients whose pain levels were moderate and low continued the incentive spirometry application. Arterial and venous oxygen saturation values and vital signs were measured and recorded at the end of the first, second and third days postoperatively on the Application Information form.
  Interventions: Procedure: Incentive Spirometry Group

INTERVENTIONS:
Procedure: Incentive Spirometry Group — The inspiration and expiration applications of incentive spirometry (IS) involved 10-20 breaths every one to two hours, depending on the tolerance of the patients.
  During the inspiration application of IS, the head of the bed was elevated to a 45° angle, and the patient was placed in a long sitting position. The patient was requested to surround and fix the IS mouthpiece well, ensuring no gap was left between the lips. The patient was told to breathe slowly and deeply, and was asked to hold their breath for 2-3 seconds, and then to breathe normally with the IS mouthpiece in his/her mouth. The patient was advised to repeat the exercise 5-10 times, and to try to cough after every 5 exercises.
  For the applied IS expiration technique applied in the study, which had not been previously encountered in literature, the patient was requested to turn the IS upside down (clockwise,180°) and to place the mouthpiece in his/her mouth and expiration application it.
  Arms: Incentive Spirometry Group

SUMMARY:
Aims and objectives: The aims of this study is to determine the effect of incentive spirometry on arterial blood gas and venous oxygen saturation and vital signs, in addition to pulmonary rehabilitation care before and after coronary artery bypass graft surgery. The objectives; were to accelerate the healing process by reducing pulmonary complications.

Background: Nurses, who carry much of the responsibility for the basic care of patients surgery play a highly important role. As a result of strong care, the recovery process of the patients will be accelerated, the hospitalization period will be shortened and morbidity and mortality will be prevented.

Design and Methods: Included in this randomized controlled study were 32 patients who underwent coronary arterial bypass graft surgery (16 in experimental group; 16 in control group) in a university hospital. Incentive spirometry is applied in the study along with an identified inspiration technique and an expiration technique that has not been previously encountered in literature. The preoperative measured values of the patients were compared with the arterial blood gas and venous oxygen saturation values and vital signs on the first, second and third postoperative days. In this study, the CONSORT checklist was followed.

DETAILED DESCRIPTION:
METHODS Design The patients in this dual-group, quasi-experimental randomized controlled study were divided into control and experimental groups using a block randomization method.

Study sample This study consisted of 32 patients (16 in the experimental group; 16 in the study group) who were hospitalized in the cardiovascular surgery clinic of a university hospital and underwent Coronary Artery Bypass Graft (CABG) surgery between December 2019 and February 2020. As a result of the power analysis using the G*Power 3.0.10 program with the data obtained from the research; the power of the study was found to be 85% for f=0.2251 effect size, 5% margin of error and n=32 sample number.

Data collection "Personal Information" and "Application Information" forms prepared by the researcher were used for the collection of data. The Personal Information Form (PIF) was prepared by the researcher after a review of previous studies, and included questions about age, body mass index (BMI), gender, chronic disease, alcohol and cigarette use, physical exercise, diet and American Society of Anesthesiologists (ASA) classification. The last preoperative arterial blood gas value, the values from the first, second and third postoperative days, as well as the venous oxygen saturation values and vital signs, were recorded on the application information form. Written informed consent was obtained from all the patients after they were explained the purpose of the study, and all took part in face-to-face interviews for the garnering of data.

Incentive Spirometry (IS) is designed to mimic the natural sighing or yawning maneuvers. The technique was used with a deep inspiration focus, as described previously in literature. Unlike in previous studies, IS was used in the present study not only for inspiration but also for expiration. In normal use, IS involves the raising of three balls side by side in transparent plastic tubes during each deep inspiration, but when turned upside down, the device can be applied also to expiration. It is thus possible to use the IS with both inspiration and expiration techniques, with positive effects on the patient in both uses. The present study made use of flow-focused IS with both the inspiration and expiration techniques, in addition to such routine clinical procedures as breathing exercises, coughing exercises, early mobilization and pain control.

The ethical aspect of the study Ethics committee approval (Date: 28.12.2017 Reference Number: 72 Decision Number: 8) was granted by the Non-Invasive Clinical Research Ethics Committee and the necessary institutional permissions were obtained from the hospital in which the research was conducted. The study was carried out in compliance with the principles of the Declaration of Helsinki, as revised in 2008. The patients included in the study were informed about the study, the aim of the study was explained, and their verbal and written consent for participation in the study was obtained.

Statistical analysis The Statistical Package for the Social Sciences (SPSS) Statistics (Version 24.0) package program was used for the statistical analyses. Frequency tables and descriptive statistics were used for the interpretation of the findings. Parametric methods were used for measurement values with a normal distribution. In accordance with parametric methods, the measurement values of two independent groups were compared with an Independent Sample t test (t-table value) and the measurement values of three or more dependent groups were compared with a Repeated Measures test (F-table value). Non-parametric methods were used for normally distributed measurement values. In accordance with non-parametric methods, the measurement values of two independent groups were compared with a Mann-Whitney U test (Z-table value) and the measurement values of three or more dependent groups were compared with a Friedman test (χ2-table value). Pearson-χ2 crossbars were used for the examination of the relationships between two qualitative variables. Consolidated Standards of Reporting Trials (CONSORT) checklist, guidelines for reporting of randomized controlled trials were used as the reporting guideline for this study.

ELIGIBILITY:
Inclusion Criteria:

* willing participants who could communicate
* with a stable clinical condition
* between 18 and 88 years old
* with no hearing problems
* with no previous psychiatric or mental illness
* undergoing coronary artery bypass surgery for the first time (non-emergency surgery)

Exclusion Criteria:

* unstable clinical situation
* declined to participate,
* history of Chronic Obstructive Pulmonary Disease (COPD) or Chronic Kidney Failure (CKD)
* those with post-operative cognitive and neurological complications and severe hemodynamic dysfunction
* those requiring resternotomy or prolonged mechanical ventilation (more than 24 hours)
* with complications (pneumonia, atelectasis , pleural effusion, etc.).

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Change from arterial blood gas parameters at 4 days | Preop, Postop 1.day, Postop 2.day, Postop 3.day
  Arterial blood gas repeated measurements were made on Preop, Postop 1.day, Postop 2.day, Postop 3.day. Among the arterial blood gas criteria, PaCO2 (35_45mmHg), Pa02 (80-100mmHg), arterial oxygen saturation (SaO2) (95-97%) values were examined. These measurements were compared between the experimental group and the control group. Measurements were made at the end of the day.
Change from venous oxygen saturation parameters at 4 days | Preop, Postop 1.day, Postop 2.day, Postop 3.day
  Venous oxygen saturation (Venous O2 /%90-100) repeated measurements were made on Preop, Postop 1.day, Postop 2.day, Postop 3.day. These measurements were compared between the experimental group and the control group. Measurements were made at the end of the day, during the resting time of the patients.
Vital signs- Change from systolic and diastolic blood pressure at 4 days (mmHg) | Preop, Postop 1.day, Postop 2.day, Postop 3.day
  In this study, systolic and diastolic blood pressure values, which are vital signs, were measured repeatedly on Preop, Postop 1.day, Postop 2.day, Postop 3.day. Measurements were made at the end of the day, during the resting time of the patients.
Vital signs- Change from respiratory rate per minute at 4 days | Preop, Postop 1.day, Postop 2.day, Postop 3.day
  In this study, respiratory rate per minute values, which are vital signs, were measured repeatedly on Preop, Postop 1.day, Postop 2.day, Postop 3.day. Measurements were made at the end of the day, during the resting time of the patients.
Vital signs- Change from heart rate per minute at 4 days | Preop, Postop 1.day, Postop 2.day, Postop 3.day
  In this study, heart rate per minute values, which are vital signs, were measured repeatedly on Preop, Postop 1.day, Postop 2.day, Postop 3.day. Measurements were made at the end of the day, during the resting time of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agostini P, Calvert R, Subramanian H, Naidu B. Is incentive spirometry effective following thoracic surgery? Interact Cardiovasc Thorac Surg. 2008 Apr;7(2):297-300. doi: 10.1510/icvts.2007.171025. Epub 2007 Nov 26. PMID 18039692
- [Background] Boden I, Skinner EH, Browning L, Reeve J, Anderson L, Hill C, Robertson IK, Story D, Denehy L. Preoperative physiotherapy for the prevention of respiratory complications after upper abdominal surgery: pragmatic, double blinded, multicentre randomised controlled trial. BMJ. 2018 Jan 24;360:j5916. doi: 10.1136/bmj.j5916. PMID 29367198
- [Background] Carvalho CR, Paisani DM, Lunardi AC. Incentive spirometry in major surgeries: a systematic review. Rev Bras Fisioter. 2011 Sep-Oct;15(5):343-50. doi: 10.1590/s1413-35552011005000025. Epub 2011 Oct 14. PMID 22002191
- [Background] Eltorai AEM, Baird GL, Eltorai AS, Healey TT, Agarwal S, Ventetuolo CE, Martin TJ, Chen J, Kazemi L, Keable CA, Diaz E, Pangborn J, Fox J, Connors K, Sellke FW, Elias JA, Daniels AH. Effect of an Incentive Spirometer Patient Reminder After Coronary Artery Bypass Grafting: A Randomized Clinical Trial. JAMA Surg. 2019 Jul 1;154(7):579-588. doi: 10.1001/jamasurg.2019.0520. PMID 30969332
- [Background] Eltorai AEM, Szabo AL, Antoci V Jr, Ventetuolo CE, Elias JA, Daniels AH, Hess DR. Clinical Effectiveness of Incentive Spirometry for the Prevention of Postoperative Pulmonary Complications. Respir Care. 2018 Mar;63(3):347-352. doi: 10.4187/respcare.05679. Epub 2017 Dec 26. PMID 29279365
- [Background] Lumb AB. Pre-operative respiratory optimisation: an expert review. Anaesthesia. 2019 Jan;74 Suppl 1:43-48. doi: 10.1111/anae.14508. PMID 30604419
- [Background] Moradian ST, Heydari AA, Mahmoudi H. What is the Role of Preoperative Breathing Exercises in Reducing Postoperative Atelectasis after CABG? Rev Recent Clin Trials. 2019;14(4):275-279. doi: 10.2174/1574887114666190710165951. PMID 31291879
- [Background] Pantel H, Hwang J, Brams D, Schnelldorfer T, Nepomnayshy D. Effect of Incentive Spirometry on Postoperative Hypoxemia and Pulmonary Complications After Bariatric Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 May 1;152(5):422-428. doi: 10.1001/jamasurg.2016.4981. PMID 28097332
- [Background] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401
- [Result] Agostini P, Singh S. Incentive spirometry following thoracic surgery: what should we be doing? Physiotherapy. 2009 Jun;95(2):76-82. doi: 10.1016/j.physio.2008.11.003. Epub 2009 Mar 3. PMID 19627688